CLINICAL TRIAL: NCT06710470
Title: Deucravacitinib Pregnancy Study: A Retrospective Observational Study on the Safety of Deucravacitinib Exposure in Pregnant Women and Their Offspring
Brief Title: A Study on the Safety of Deucravacitinib Exposure in Pregnant Women and Their Offspring
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM011-201
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — deucravacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Cohort 1: Participants exposed to deucravacitinib for the full pregnancy duration
  Interventions: Drug: Deucravacitinib
- Cohort 2: Participants exposed to deucravacitinib for the first trimester
  Interventions: Drug: Deucravacitinib
- Cohort 3: Participants exposed to deucravacitinib for the first 20 weeks of gestation
  Interventions: Drug: Deucravacitinib
- Cohort 4: Participants exposed to other systemic psoriasis medications for the full pregnancy duration
  Interventions: Drug: Systemic psoriasis medications
- Cohort 5: Participants exposed to other systemic psoriasis medications for the first trimester
  Interventions: Drug: Systemic psoriasis medications
- Cohort 6: Participants exposed to other systemic psoriasis medications for the first 20 weeks of gestation
  Interventions: Drug: Systemic psoriasis medications
- Cohort 7: Participants not exposed to any systemic medications for the full pregnancy duration
  Interventions: Other: No systemic medications
- Cohort 8: Participants not exposed to any systemic medications during the first trimester
  Interventions: Other: No systemic medications
- Cohort 9: Participants not exposed to any systemic medications during the first 20 weeks of gestation
  Interventions: Other: No systemic medications

INTERVENTIONS:
Drug: Deucravacitinib — As per product label
  Groups: Cohort 1; Cohort 2; Cohort 3
Drug: Systemic psoriasis medications — As per product label
  Groups: Cohort 4; Cohort 5; Cohort 6
Other: No systemic medications — Participants not exposed to any systemic medications
  Groups: Cohort 7; Cohort 8; Cohort 9

SUMMARY:
This observational study aims to assess pregnancy and infant outcomes among pregnant women with psoriasis who have been exposed to deucravacitinib treatment in the USA.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age 15 through 50 years at date of conception
* Start of pregnancy, defined as the estimated date of conception, during the accrual period (09-Sep-2022 through 31-Oct-2026)
* Continuous medical and pharmacy coverage for a minimum of 6 months prior to and including the estimated date of conception
* Presence of psoriasis from 12 months prior to the date of conception through the end of pregnancy

Exclusion Criteria:

• Exposure to any known teratogens from 5 half-lives prior to the estimated date of conception through the end of the relevant exposure window

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will include women aged 15 through 50 years with psoriasis who become pregnant (based on their estimated date of conception) from 09-Sep-2022 through 31-Oct-2026 that have been identified in the Optum Research Database (ORD).
Sampling Method: Non-Probability Sample
Enrollment: 833 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of infants born with Major Congenital Malformations (MCMs) | Up to 12 months after birth or date of health plan disenrollment
  MCMs defined as a structural abnormality with surgical, medical, or cosmetic importance (excluding chromosomal abnormalities or physiological features due to complications of prematurity, such as cryptorchidism, inguinal hernia, or isolated patent ductus arteriosus in infants born less than 37 weeks of gestation)

SECONDARY OUTCOMES:
Pregnancy outcomes | Up to 9 months or date of health plan disenrollment
  Incidence of the following pregnancy outcomes: spontaneous abortion, induced abortion, ectopic pregnancy, stillbirth, pre-eclampsia, eclampsia and gestational diabetes
Infant outcomes | Up to 12 months after birth or date of health plan disenrollment
  Incidence of the following infant outcomes: small for gestational age, large for gestational age, low birthweight, preterm birth, serious or opportunistic infections, postnatal growth deficiency, infant developmental deficiency, neonatal hospitalization, and infant/neonatal/perinatal death

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Bristol-Meyers Squibb, Lawrenceville, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts